CLINICAL TRIAL: NCT06922864
Title: the Prediction Value of Combined Electroencephalographic and Electromyographic Response in Disorders of Consciousness
Status: Not yet recruiting | Type: Observational
Sponsor: KY20242235jiangwen (Other)
Responsible Party: Sponsor-Investigator, KY20242235jiangwen, head of department, Xijing Hospital
Organization: Xijing Hospital (Other)
Other Study IDs: KY20242235jiangwen
Record Dates: First submitted 2025-04-03; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Disorders of Consciousness Due to Severe Brain Injury
MeSH Terms: interventions — UBE3A protein, human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- good outcome
- not good outcome

INTERVENTIONS:
Other: thermal stimulation — contact heat stimulation at 54℃
Other: itch — itch the sole of the foot

SUMMARY:
The goal of this observation study is to learn about the prediction value of combined electroencephalographic and electromyographic response in disorders of consciousness.

The main ways of stimulation is thermal and itch. Six months after inclusion in the study, patients were classified according to the Glasgow Outcome Scale Extended, (GOSE).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Brain damage lasts 28 to 90 days.
3. It meets the diagnostic criteria of unresponsive arousal syndrome/vegetative state (UWS/VS) or microconscious state (MCS).

   Diagnostic criteria for UWS/VS: loss of cognitive function and inability to execute commands; There is a sleep-wake cycle; Inability to understand or express language; The ability to open eyes automatically or in response to stimulation; Can be purposeless eye following movement; The functions of hypothalamus and brainstem were basically preserved.

   MCS diagnostic criteria: simple instructions can be executed; Yes/no (whether correct or not) can be expressed by gesture or speech; Have an understandable language; Purposeful behavior (including activity or emotional response) with more than one can diagnose MCS.
4. All subjects' legal guardians sign informed consent forms.

Exclusion Criteria:

1. Spinal cord T1 and above plane injury, peripheral nerve injury and so on affect nerve conduction;
2. The impact of injury on palms and soles of feet;
3. History of developmental, psychiatric, or neurological disorders prior to brain injury.
4. Deep sedation within 72 hours, including the use of general anesthesia.
5. Increased intracranial pressure, liver/kidney failure, and hemodynamic instability within 72 hours.
6. Severe co-existing systemic diseases with limited life expectancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients wih disorders of consciousness in xijing hospital
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
the state of consciousness | 6 months

SECONDARY OUTCOMES:
the score of GOSE | 6 months